CLINICAL TRIAL: NCT06183957
Title: The Effect of Shower on Birth Pain, Postpartum Fatigue and Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Ayca Solt Kirca, Asssociate professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KırklareliAS-9
Record Dates: First submitted 2023-12-12; First posted 2023-12-28 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Pain; Fatigue
Keywords: Postpartum period; Postpartum comfort; Hydrotherapy
MeSH Terms: conditions — Pain; Fatigue

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydrotherapy group (Experimental): When women in this group are taken to their labor rooms (when the dilation is 4-5cm), they should be standing or standing, depending on their preferences, on their waist, abdomen or whole body, with the temperature of the water between 32-37 °C (the temperature preferred by the woman will be applied) for at least 20 minutes. Sitting shower application will be performed under the observation of the researcher midwife. The temperature of the flowing water will be measured with a bucket and a thermometer that helps evaluate the temperature. The application will be repeated when the dilation is 6-8 cm.
  Interventions: Other: hydrotherapy group
- Control group (No Intervention): Women in this group will not undergo any treatment other than routine hospital protocol (midwifery care). Additionally, the vital signs (blood pressure, pulse) of the participants will be measured and recorded hourly by the midwife. These data will be recorded in each participant's file.

INTERVENTIONS:
Other: hydrotherapy group — When women in this group are taken to their labor rooms (when the dilation is 4-5cm), they should be standing or standing, depending on their preferences, on their waist, abdomen or whole body, with the temperature of the water between 32-37 °C (the temperature preferred by the woman will be applied) for at least 20 minutes. Sitting shower application will be performed under the observation of the researcher midwife. The temperature of the flowing water will be measured with a bucket and a thermometer that helps evaluate the temperature. The application will be repeated when the dilation is 6-8 cm.
  Arms: hydrotherapy group

SUMMARY:
According to the definition of the International Association for the Study of Pain, pain; It is an unpleasant sensory and emotional sensation and behavior related to the individual's past experiences, caused by real or potential tissue damage originating from any part of the body. Birth pain is the most severe pain experience known and defined, with physiological as well as psychological and sociocultural components that may vary among individuals.Pharmacological and non-pharmacological applications are used to relieve birth pain. While pharmacological methods reduce pain, they distract women from the physiological reality of birth and prevent women from accepting pain as a natural part of birth. Non-pharmacological methods are alternative options that will help women manage pain during birth by ensuring that women experience pain.

Showering (hydrotherapy), one of the non-pharmacological methods used to reduce pain in labor, is used to increase relaxation and reduce birth pain. In a study conducted domestically, it was stated that the use of hydrotherapy during labor pain helped the woman relax, reduced the pain felt, lowered blood pressure and increased diuresis. Fatigue, in addition to being a universal symptom associated with diseases, is also a common complaint among healthy individuals.

In line with the literature information, this study aims to examine the effect of shower applied during birth on postpartum fatigue and postpartum comfort.

DETAILED DESCRIPTION:
According to the definition of the International Association for the Study of Pain, pain; It is an unpleasant sensory and emotional sensation and behavior related to the individual's past experiences, caused by real or potential tissue damage originating from any part of the body. Birth pain is the most severe pain experience known and defined, with physiological as well as psychological and sociocultural components that may vary among individuals. Physiological components; The pressure on the tissues of the birth canal and the stretching of the tissues are psychosocial components; It is related to fear, anxiety and coping ability during the birth process. The individual's response to pain with cultural values and learned behaviors constitutes the sociocultural dimension of pain. In addition to these known characteristics of labor pain, the degree of pain varies according to the frequency, duration and intensity of contractions and the cervical opening. The American Society of Obstetrics and Gynecology states that labor pain should be treated and that it may have negative effects on maternal and neonatal health in cases where the pregnant woman has difficulty coping with labor pain.

Pharmacological and non-pharmacological applications are used to relieve birth pain. While pharmacological methods reduce pain, they distract women from the physiological reality of birth and prevent women from accepting pain as a natural part of birth. Non-pharmacological methods are alternative options that will help women manage pain during birth by ensuring that women experience pain. The World Health Organization (WHO) recommends the use of non-pharmacological methods such as massage and touching, distraction and imagination, movement and position, music, making sounds and praying, aromatherapy, hydrotherapy, acupressure, hot and cold applications in labor pain.

Showering (hydrotherapy), one of the non-pharmacological methods used to reduce pain in labor, is used to increase relaxation and reduce birth pain. In a study conducted domestically, it was stated that the use of hydrotherapy during labor pain helped the woman relax, reduced the pain felt, lowered blood pressure and increased diuresis. The use of water during labor and regular feeding of the uterus in the first stage of labor has helped to feel less pain during contractions and to have shorter and less invasive births.

Fatigue, in addition to being a universal symptom associated with diseases, is also a common complaint among healthy individuals. The North American Nursing Diagnosis Association (NANDA) defines fatigue as "a predominant, persistent feeling of exhaustion and a decrease in normal physical and mental working capacity". defines. Symptoms of fatigue; Inability to carry out daily tasks, impaired concentration, difficulty in remembering, short-term memory loss, indifference to the environment, decreased awareness, lack of energy, fatigue, difficulty in making decisions, muscle weakness, increased physical complaints, emotional changes, tendency to sleep, hallucinations, perceptual weakness. is suffering.

Fatigue is a common symptom during pregnancy, birth and the postpartum period. In addition to being a very special, happy experience for women, birth also means coping with physical pain and difficulties and fatigue due to insomnia. With the birth, the six-week period begins, called the postpartum period, during which the woman feels social, physical and psychological changes. This process is a woman's; It is a difficult period in which all systems and organs in the body return to their pre-pregnancy state, the woman tries to adapt to the new roles and responsibilities acquired in the transition to parenthood, and many progressive and regressive changes occur in the woman's body. Fatigue, which is an inevitable part of this period, can increase until the sixth postpartum week. In the study of Kılıç et al., it was reported that 88.5% of women experienced fatigue in the postpartum period.

In line with the literature information, this study aims to examine the effect of shower applied during birth on postpartum fatigue and postpartum comfort.

ELIGIBILITY:
Inclusion Criteria:

* -Voluntarily agreeing to participate in the study
* She will have her second birth spontaneously vaginally at term (between 37-42 weeks of pregnancy).
* The fetal weight estimated by ultrasound is 2500-4000 grams
* Single fetus and head presentation
* Being in the active phase of labor (cervical dilation 4 cm)
* Ability to establish written/verbal communication
* Not taking any analgesia or anesthesia to relieve pain and fatigue before birth and during labor.
* Newborn APGAR score is 7 or above

Exclusion Criteria:

* giving up on research
* Having received infertility treatment
* Birth by cesarean section
* Having an interventional birth (forceps, vacuum, episiotomy application)
* Being primiparous, having a third or more birth (grandmultiparous)
* Having any systemic, chronic and neurological disease (Diabetes Mellitus, Hypertension, Thyroid diseases, Multiple Sclerosis, Epilepsy, etc.)
* Regular use of medication due to any disease
* Receiving psychiatric treatment (pharmacotherapy/psychotherapy)
* Any induction application that will affect uterine contractions and dilation
* Having any pregnancy complications (placenta previa, preeclampsia, premature rupture of membranes, oligohydramnios and polyhydramnios, contraction anomalies, presentation disorder, intrauterine growth retardation, intrauterine dead fetus, macrosomic babies, fetal distress, etc.)
* Having any problem that prevents communication (such as not knowing Turkish, hearing, speaking and understanding impairment),

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 80 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | 1 week
  sociodemographic characteristics, medical and obstetric pregnancy history, the woman's current pregnancy, prenatal and postpartum period

SECONDARY OUTCOMES:
Visual Comparison Scale (VAS) | during labour period (up to 10 hours)
  It is stated that the Visual Comparison Scale (VAS) is more sensitive and reliable in measuring pain intensity than other unidimensional scales. VAS is a 10 cm ruler with no pain written on one end and the most severe pain possible on the other end. Evaluation of VAS is defined as No pain: 0 cm, Mild pain: 0.5 cm - 3.0 cm, Moderate pain: 3.5 cm - 6.5 cm, Severe pain: 7.0 cm - 10.0 cm. VAS is a very sensitive method in the evaluation of pharmacological and non-pharmacological treatments that reduce pain and is a scale in the form of vertical or horizontal, visual, numerical or descriptive analogue.
Postpartum Comfort Scale (WSCO) | between 2-4 hours postpartum period
  It is a scale that can be used appropriately and safely in measuring the postpartum comfort of mothers who have given birth by normal birth or cesarean section, in meeting postpartum comfort needs, and in evaluating the outcome as a concrete indicator of the outcome. Its consists of 34 items. A 5-point Likert-type scale scoring system was used to enable an evaluation for each item that determines the situation to be measured. For each item, expressions and scoring ranging from "completely agree" (5 points) to "strongly disagree" (1 point) were made. The lowest score to be obtained from the scale is 34 and the highest score is 170.
Person-Oriented Maternity Care Scale | between 2-4 hours postpartum period
  The original scale has 30 items and 3 subscales. The Turkish form consists of 21 items and 3 sub-dimensions. Except for items 6, 11 and 13 (5 options and coded as 0, 1, 2, 3, 4), the remaining items have 4 options ("no, never" 0, "yes, a few times" 1, "yes, most of the time" "time" is scored as 2, "yes, always" is scored as 3). The lowest score that can be obtained from the total scale is 0, the highest score is 66, the lowest score that can be obtained from the "Value and Respectful Care" sub-dimension (2,3,4,5) is 0, the highest score is 12, "Communication and Autonomy" (1,6,7). The lowest score that can be obtained from the "Supportive Care" sub-dimension (12,13,15,16,17,18,19,20,21) is 0 and the highest score is 26. The lowest score is 0 and the highest score is 28. As the score increases, mother-focused care increases.

CONTACTS AND LOCATIONS:
Overall Officials: ZEYNEP CAMBAZ, Principal Investigator — Tekirdağ Çorlu İlçe Devlet Hastanesi
Locations (1):
- Tekirdağ Çorlu District State Hospital, Tekirdağ, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No